CLINICAL TRIAL: NCT06351501
Title: Evaluation of the Effectiveness of Hormonal Treatment in Adolescents Suffering from Gender Dysphoria
Acronym: TRANSADO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P170923J; 2019-000300-16 (EudraCT Number)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Gender Dysphoria
Keywords: Gender Dysphoria; adolescents; hormonal treatment; mental health
MeSH Terms: conditions — Gender Dysphoria; Psychological Well-Being | interventions — Testosterone

STUDY DESIGN:
Intervention Model Description: Multicenter, controlled, randomized, open trial with blinded evaluation of the primary endpoint (Prospective Open Blinding Endpoint PROBE study). Randomization will be stratified by sex assigned at birth and the investigating center. The primary analysis will be intention-to-treat and multiple imputation methods will be used to handle missing data. After verification of the inclusion criteria by the child psychiatrist (selection visit), then the pediatric endocrinologist (inclusion visit), the adolescent will be included in the study and will benefit from an initial evaluation (T0) by a psychologist trained for the primary criterion (CGAS) and secondary psycho-affective criteria. The patients will then be sent again to the pediatric endocrinologist who will randomize the patient (via an IT platform) and give them the treatment corresponding to their assigned group.
Who Masked: Outcomes Assessor
Masking Description: The assessment of the primary criteria will be carried out by a psychologist who will have no knowledge of the teenager's allocation group and will not have been involved in his or her care. At T1, the assessment will be based on key elements of the patient's file provided to him or her without any element that could indicate his or her allocation group or original gender, and a telephone interview with the teenager and his or her parents in which they will have been told in advance not to reveal the allocation group or gender. The psychologist who assesses a 16-year-old will be different from the one who assesses a 14-year-old. Psychological assessments other than the primary criterion, and the assessment by the pediatric endocrinologist, will take place at the site of the patient's usual care. Adolescents will be monitored as part of their usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- early hormonal treatment (Experimental): early hormonal treatment initiated at 14 years +/- 6 months, in addition to usual care
  Interventions: Drug: hormonal treatment with cross sex hormones (testosterone or oestrogenes) started at 14 years old +/- 6 months
- usual treatment (Active Comparator): Usual care between 14 and 16 years +/- 6 months : child psychiatric consultations, endocrinological consultations and consultations with a psychologist, family interviews, network work with local health partners and national education.
  Then hormonal treatment initiated at 16 years +/- 6 months, in addition to usual care.
  Interventions: Drug: Cross sex hormones ( œstrogenes or testosterone) started at 16 years old +/- 6 months

INTERVENTIONS:
Drug: hormonal treatment with cross sex hormones (testosterone or oestrogenes) started at 14 years old +/- 6 months — 4 years of follow up (FU) with evaluation at T0 (14 years old +/- 6 months), T1 (16 years old +/-6 months) and T2 (18 years old+/- 6 months) with eather ANDROGEL® 16.2 mg/g, gel (testostérone) or ESTREVA® 0.1 %, gel ou 1.3 PROVAMES® 1 mg, cp (oestrogenes)
  Arms: early hormonal treatment
Drug: Cross sex hormones ( œstrogenes or testosterone) started at 16 years old +/- 6 months — 2 years of hormonal treatment from 16 old +/- 6 months to 18 years old +/- 6 months
  Arms: usual treatment

SUMMARY:
Gender dysphoria (GD) is a significant suffering lasting more than 6 months in a subject, with regard to the discrepancy felt between his or her gender identity and his or her birth sex. From the onset of puberty, most of these self-identified transgender adolescents will persist in their transgender identity and will undergo hormonal and surgical reassignment when the time comes. International best practice guidelines recommend early treatment from the start of pubertal development to block pubertal progression, with the possibility of hormonal transition by administering sex hormones of the desired sex usually around the age of 16. However, in order to reduce the psychosocial consequences of GD, more and more referral teams are carrying out this transition from the age of 14, although no study has been published to show its benefit compared with a transition at the age of 16. In the absence of treatment, co-morbidity among adolescents suffering from gender dysphoria is very high, with anxiety-depressive states, suicidal risk and dropping out of school in the forefront. Our hypothesis is that hormonal transition started at an age closer to physiological puberty can significantly reduce this comorbidity and improve quality of life for these adolescents. This is the first therapeutic trial to be conducted in France in the transgender adolescent population, in an area where international recommendations based on the principles of Evidence Based Medicine are essentially derived from the clinical expertise of teams who have specialized in the care of transgender people for over forty years, while clinical data derived from structured research are still very scarce.

The results of this study will guide the care of transgender adolescents, allowing them, if the study is positive, to access hormonal treatments earlier and thus more quickly improve their overall functioning, anxiety-depressive symptoms and their quality of life.

DETAILED DESCRIPTION:
Multicenter, controlled, randomized, open trial with blinded evaluation of the primary endpoint (Prospective Open Blinding Endpoint PROBE study). Randomization will be stratified by sex assigned at birth and the investigating center. The primary analysis will be intention-to-treat and multiple imputation methods will be used to handle missing data. After verification of the inclusion criteria by the child psychiatrist (selection visit), then the pediatric endocrinologist (inclusion visit), the adolescent will be included in the study and will benefit from an initial evaluation (T0) by a psychologist trained for the primary criterion (CGAS) and secondary psycho-affective criteria.The patients will then be sent again to the pediatric endocrinologist who will randomize the patient (via an IT platform) and give them the treatment corresponding to their assigned group. Adolescents in both groups will be reassessed at 16 years +/- 6 months (T1). At the end of this evaluation, patients in the control group will begin their hormonal treatment. Adolescents will undergo a final evaluation at 18 years +/- 6 months (T2), at which time the same criteria as at T0 and T1 will be collected.

Main objective: To evaluate, in gender dysphoric adolescents, having completed their social transition, having or not undergone prior pubertal suppression, the effectiveness of hormonal treatment with estrogens or testosterone initiated at 14 years +/- 6 months of age on the overall functioning of the teenager at 16 years +/- 6 months old.

Primary endpoint: Children's Global Assesment Scale (CGAS) score at age 16 +/- 6 months

Secondary objectives : Evaluate, in gender dysphoric adolescents who have completed their social transition, whether or not they have benefited from prior pubertal suppression:

* the effectiveness of hormonal treatment started at 14 years old +/- 6 months vs. 16 years old +/- 6 months on the overall functioning of the adolescent at 18 years old+/- 6 months,
* the safety (side effects) of hormonal treatment started at age 14 +/- 6 months,
* and the relevance of hormonal treatment started at 14 years old +/- 6 months on other parameters assessed at 16 +/- 6 months and 18 +/- 6 months years old (gender identity, depression, anxiety, emotional, behavioral disorders and other comorbidities, objective and subjective quality of life, body image, height, waist/hip ratio, bone mineral density, BMI).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 14+/- 6 months,
* Having initiated puberty: tanner score ≥2 for FtM; tanner score ≥2 (clinic and/or testosterone >0.3 ng/mL) for MtF
* Presenting the criteria for gender dysphoria according to the DSM5 assessed by at least two child psychiatric interviews at least six months apart where the diagnosis of gender dysphoria was clinically established and that of associated autism spectrum disorder refuted and/or associated cognitive impairment, confirmed by specific scales (Gender Identity / Gender Dysphoria Questionnaire for Adults and Adolescents (GIDYQ-AA) and Utrecht Gender Dysphoria Scale (UGDS))
* Whose indication for hormonal transition has been validated in a multidisciplinary consultation meeting after at least one consultation with the pediatric endocrinologist with clinical examination, blood pressure measurement, and information on hormonal treatments in the context of gender dysphoria.

Exclusion Criteria:

* Contraindication to hormonal treatment (see paragraph 1.5)
* Hormonal treatment needs to be adjusted (FtM patients treated with anti-coagulants or with thrombophilia).
* Patients with risk of aggravation of certain diseases under oestrogen treatment (MtF patients with uncontrolled diabetes with HBA1C > 8%, patients with cholelithiasis, biliary lithiasis, systemic lupus erythematosus, severe asthma, severe arterial hypertension, severe migraines, otosclerosis, epilepsy not controlled by treatment).
* Patients with cancer with a risk of hypercalcemia (and associated hypercalciuria), linked to bone metastases.
* Severe cardiac, hepatic or renal failure or ischemic heart disease, due to the risk of severe complications characterized by edema, with or without congestive heart failure.
* Uncontrolled high blood pressure.
* Patients with epilepsy and migraine.
* Patients with current or history of thromboembolic events.
* Severe untreated chronic depression
* Current anticoagulant treatment
* Severe autism Spectrum Disorder (clinical screening, confirmed in cases of doubt by the Social Responsiveness Scale (SRS) Raw-score > 76, carried out as part of usual care in cases of clinical evidence,
* Cognitive deficit (clinical screening, confirmed by an QI < 80 on the Weschler scale (WISC V), carried out as part of the usual treatment in the event of clinical evidence.
* Refusal to participate in the study on the part of the adolescent or one of the holders of parental authority (both holders and the adolescent must sign a written consent after receiving appropriate information).
* No social security cover
* Participation in other intervention research
* Pregnancy in progress
* Insufficient knowledge of French

Ages: 162 Months to 174 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2029-06-24 (Estimated); Study Completion 2031-06-24 (Estimated)

PRIMARY OUTCOMES:
Global functionning using the Children's Global Assessment Scale (CGAS) | 16 years old +/- 6 months
  The Children's Global Assessment Scale (CGAS), adapted from the Global Assessment Scale for adults, is a rating of general functioning for children and young people until 16 years old. The clinician assesses a range of aspects of psychological and social functioning and gives the child or young person a single score between 1 and 100, based on their lowest level of functioning. The score puts them in one of ten categories that range from "needs constant supervision" (1-10) to "superior functioning" (91-100). The measure can be used by clinicians as well as researchers to complement other scales measuring more specific symptoms.

SECONDARY OUTCOMES:
Drug use (DEP-ADO) | T0 (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  Drug use: assessed by specific questions via the DEP-ADO questionnaire (screening grid for problem substance use among adolescents).
  Dep-Ado is a 15 minutes questionnaire to evaluate alcohol and substance use adolescent population aged 12 to 17 years. No problem if total score <12; warning of >12 et <19; pathological use needing intervention if >20
WISC-V (weschler Test) | T0 (14 years old +/-6 months); T2 ( 18 years old +/-6 months)
  cognitive test with 4 subscales (verbal comprehension index, perceptual reasoning index, logical score, working memory index, processing speed index). IQ is calculated. If <80, it is an non inclusion criteria. Normal range between 80 and 120. when > 120 précocity
UGDS (Utrecht Gender Dysphoria Scale ) and GIDYQ-AA (Gender Identity/ Gender Dysphoria Questionnaire for Adolescents and Adults scale ) | selection visit ; T1 (16 years old +/-6 months) ; T2 (18 years old +/-6 months)
  The Utrecht Gender Dysphoria Scale (UGDS) is a validated, 12-item screening measure for both adults and adolescents used extensively in gender clinics to assess gender dysphoria. Minimal score= 12; max=60. two versions (AFAB, AMAB)
Beck Depression Inventory (BDI) | T0 (14 years old +/-6 mois); T1 (16 years old+/-6 monhs); T2 ( 18 years old +/-6 months)
  is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.Min = 0 Max = 39 Between 0 and 3 = no Dépression
Body Image Scale (BIS) | T0 (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  The 10-item BIS was developed to assess changes in body image assessed with a four-point scale from "not at all" to "very much." High scores indicate higher body image.(Min=30, Max=150 )
State and Anxiety Inventory for Children (STAI-C) | T0 (14 years old +/-6 mois); T1 (16 years old+/-6 monhs); T2 ( 18 years old +/-6 months)
  STAI-C includes 20-items that describe anxiety experiences a person might experience (e.g., item 6-"I worry too much"©). For each item, participants choose one of three options that indicate how often they experience the described situation - "hardly-ever", "sometimes" or "often"; these options are scored with 1, 2, and 3 points, respectively (total score range: 20-60). Higher scores indicate higher anxiety
World Health Organization Quality Of Life - BREF (WHOQOL-BREF) | T0 (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  This 26-item instrument measures four fields, i.e. physical health, mental health, social relations and the environment. The analysis is based on the scores generated for each field (no overall score can be calculated). The user manual is comprehensive, which makes the instrument easy to use (WHO, 1996). While some studies call into question the construct validity (D'Abundo et al., 2011), the WHOQOL-BREF is generally recognized as a reliable, valid instrument to assess quality of life and is widely used in the literature for clinical and population-based surveys (Oliveira, Carvalho and Esteves, 2016; Skevington, Lotfy and O'Connell, 2004).
Satisfaction With Life Scale (SWLS) | T0 (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  The SWLS is a short 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life. The scale usually requires only about one minute of a respondent's time.Min=5, Max=35. The higher score means a greater satisfaction with life
Height, bone mineral density, BMI, waist to hip ratio | inclusion visit (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  MI is a measurement of a person's leanness or corpulence based on their height and weight, and is intended to quantify tissue mass
Mini International Neuropsychiatric Interview (MINI) | selection visit ; T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  To assess the 17 most common psychiatric disorders and suicidality in DSM-III-R, DSM-IV and DSM-5 and ICD-10. The MINI was designed as a brief structured diagnostic interview to meet the need for a short but accurate structured psychiatric interview for multicenter clinical trials and epidemiology studies and to be used as a first step in outcome tracking in nonresearch clinical settings.
The emotional and sexual relationship | T0 (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  The emotional and sexual relationship assessed by specific questions
School drop-out / family breakdown | T0 (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  School drop-out / family breakdown assessed by specific questions
Global Assesment Scale (GAS) | T2 : 18 years old +/-6 months
  assess the adolescent's overall functioning, heteroquestionnaire, score from 1 to 100, on file and after 30-minute interview
Potential side-effects | T0 (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
Child Behaviour Checklist (CBCL) scale | T0 (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  Emotional disorders and possible comorbidities assessed by the Child Behavior Checklist (CBCL) score, parent self-questionnaire, 15 minutes
Youth Self Report (YSR) scale | T0 (14 years old +/-6 months); T1 (16 years old+/-6 months); T2 ( 18 years old +/-6 months)
  Emotional disorders and possible comorbidities: assessed by the Youth Self Report (YSR) self-questionnaire, 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: David COHEN, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Service de psychiatrie de l'enfant et de l'adolescent, GH Pitié-Salpêtrière, Paris, Paris
  - Service d'Endocrinologie et Diabétologie Pédiatrique, CHU Robert Debré, Paris, Paris
  - Service de Psychiatrie de l'enfant et de l'adolescent, CHU Robert Debré, Paris, Paris
  - Service Endocrinologie et Diabète de l'enfant, CHU Le Kremlin Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No